CLINICAL TRIAL: NCT01956864
Title: A Phase I Study of High-Dose Oral Vitamin D for the Prevention of Hepatocellular Carcinoma in Subjects With Cirrhosis
Brief Title: Study of High-Dose Oral Vitamin D for the Prevention of Liver Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI transferred from Georgetown to Johns Hopkins University. No participants enrolled at either site. Funding lapsed.
Sponsor: Johns Hopkins University (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB00047888
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
Keywords: Vitamin D
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose VD 1 (Experimental): Vitamin D
  Interventions: Drug: Vitamin D
- Dose VD 2 (Experimental): Vitamin D
  Interventions: Drug: Vitamin D
- Dose VD 3 (Experimental): Vitamin D
  Interventions: Drug: Vitamin D
- Dose VD 4 (Experimental): Vitamin D
  Interventions: Drug: Vitamin D
- Dose VD 5 (Experimental): Vitamin D
  Interventions: Drug: Vitamin D
- VD 6 Month Treatment (Experimental): Vitamin D
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Doses of vitamin D will be increased from a baseline dose to the maximum tolerated dose. There could therefore be up to 5 possible doses of Vitamin D. Once the maximum tolerated dose of vitamin D has been determined, patients will follow a regimen on that dose for 6 months.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a high dose of vitamin D (VD) in patients with cirrhosis. The investigator hypothesizes that high dose VD will be safe and well-tolerated in adults with cirrhosis, and will inhibit the inflammatory and proliferative events that cause progression of cirrhosis to hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study will be done in two phases. The first phase is being done to find the highest dose of VD that can be tolerated, in other words taken without causing severe side effects. The second phase is a 6 month treatment with the dose determined to be safe in the first phase, to investigate general health benefits and the potential to reduce the development of Hepatocellular carcinoma (HCC), also known as liver cancer. Improvement of general health will be determined by interviews with patients, markers in the blood for response to VD, bone remodeling, inflammation, and evidence of HCC on routine imaging.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects between the ages of 18 and 75 with cirrhosis of any etiology followed at the Georgetown Transplant Institute, Washington, DC, will be offered entry into this study. The diagnosis of cirrhosis will be based on clinical, imaging or histological studies.
2. No evidence of HCC on entry imaging study ( if liver nodules are present, these should be classified as LIRADS 1-3 only).
3. Model for End Stage Liver Disease (MELD) score under 22 (a MELD score over 22 would predict a 3 month mortality rate of approximately 20%).
4. Not currently participating in another intervention study.
5. Not pregnant or lactating, and willing to use effective contraception during study period.
6. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
7. Ability to provide written informed consent according to national/local regulations

Exclusion Criteria:

1. Any diagnosis of kidney stones
2. A diagnosis of granulomatous diseases (e.g., sarcoidosis), active chronic fungal or mycobacterial infections (e.g., tuberculosis, histoplasmosis, coccidioidomycosis, blastomycosis, berylliosis, or Wegener's granulomatosis) in the past 6 months
3. A diagnosis of hyperparathyroidism or other serious disturbance of calcium metabolism in the past 5 years
4. A diagnosis of severe kidney disease, e.g., chronic renal failure, in the past 6 months
5. A diagnosis of unexplained hypercalcemia in the past 6 months
6. Any diagnosis of osteoporosis with physician recommendation for treatment of low bone mass
7. A diagnosis of two or more low trauma fractures in the past 6 months
8. A diagnosis of a medical condition requiring treatment with VD (e.g., osteomalacia) in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-02-11 (Actual)

PRIMARY OUTCOMES:
Number of participants on high dose Vitamin D with adverse events | after 1 year

SECONDARY OUTCOMES:
Changes in the expression of serum and imaging biomarkers | After 6 months on vitamin D regimen

CONTACTS AND LOCATIONS:
Overall Officials: Kirti Shetty, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sibley Memorial Hospital /Johns Hopkins University, Washington D.C., District of Columbia, United States